CLINICAL TRIAL: NCT03942250
Title: Uses of Irradiated Human Amniotic Membrane in the Treatment of Dystrophic Epidermolysis Bullosa Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Atomic Energy Authority (Other Government)
Collaborators: Waleed Nemr,Egyptian Atomic Energy Authority (Unknown)
Responsible Party: Principal Investigator, Nashwa Radwan, Head of amniotic tissue laboratory, Principal Investigator, Egyptian Atomic Energy Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2222018NCRRT
Record Dates: First submitted 2018-02-22; First posted 2019-05-08 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Epidermolysis Bullosa; Chronic Skin Ulcer
Keywords: Epidermolysis Bullosa; Amniotic membrane
MeSH Terms: conditions — Epidermolysis Bullosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated (Experimental): Patients who received REGE pro dressing on EB wounds lesion weekly for 10 weeks
  Interventions: Biological: REGE pro dressing

INTERVENTIONS:
Biological: REGE pro dressing — REGE pro is a dressing of dried human amniotic membrane sterilized by gamma radiation

SUMMARY:
To evaluate the effect of human amniotic membrane as a weekly dressing on chronic wounds in Epidermolysis Bullosa (EB) patients.

DETAILED DESCRIPTION:
Dried human amniotic membrane dressing were obtained from National center for radiation research and technology, Egypt (NCRRT), under commercial name REGE pro.

ELIGIBILITY:
Inclusion Criteria:

1- Patients diagnosed as EB wounds must be chronic

Exclusion Criteria:

1. Patients Must stop other line of treatment
2. Exclude patients have:

   1. Autoimmune diseases
   2. Diabetes

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Lesion area | 6 weeks
  The lesion area from the first treatment is greater than 2 cm^2 (grade 3, according to CTCAE v4.0), to the complete healing (= 0 cm^2).
Clinical progression sings | 6 weeks
  * After the first application time: White transperent color of granulation tissue appeared.
  * After the second application time: color dense of granulation tissue increased and covered all over the wound.
  * After the third application time: granulation tissue thickness increased and appeared as a complete homogenous layer.
  * After the fourth application time: depending on lesion depth and size, granulation tissue turned to be pink to red color.
  * After the fifth and sexth application time: Skin layers development appeared.

SECONDARY OUTCOMES:
Patient complain (upon the weekly questionnaire) | 6 weeks
  The quality of life is scored 0 (minimum) -100 (maximum), the pain reduction is scored 0-100 (as previous) from the first visit till 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Nashwa K Radwan, PhD, Study Director — NATIONAL CENTER FOR RADIATION RESEARCH AND TECHNOLOGY
Locations (1):
- Amniotic tissue lab, Cairo, Egypt

REFERENCES:
- [Background] Nemr W, Bashandy AS, Araby E, Khamiss O. Biological Activity Alterations of Human Amniotic Membrane Pre and Post Irradiation Tissue Banking. Pak J Biol Sci. 2016;19(7):289-298. doi: 10.3923/pjbs.2016.289.298. PMID 29023030
- [Result] Lo V, Lara-Corrales I, Stuparich A, Pope E. Amniotic membrane grafting in patients with epidermolysis bullosa with chronic wounds. J Am Acad Dermatol. 2010 Jun;62(6):1038-44. doi: 10.1016/j.jaad.2009.02.048. PMID 20466177